CLINICAL TRIAL: NCT02853344
Title: A Phase II Single-arm, Open-label Monotherapy Clinical Trial of Pembrolizumab (MK-3475) in Locally Advanced/Metastatic Renal Cell Carcinoma (mRCC) (KEYNOTE-427)
Brief Title: Study of Pembrolizumab (MK-3475) Monotherapy in Locally Advanced/Metastatic Renal Cell Carcinoma (MK-3475-427/KEYNOTE-427)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-427; MK-3475-427 (Other: Merck Protocol Number); 2016-000589-47 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Clear Cell RCC (Experimental): Participants with clear cell RCC receive pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 doses (approximately 24 months).
  Interventions: Biological: Pembrolizumab
- Cohort B: Non-clear Cell RCC (Experimental): Participants with non-clear cell RCC receive pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The purpose of this study is to assess the safety and efficacy of monotherapy pembrolizumab (MK-3475) in participants with renal cell carcinoma (RCC). There will be two cohorts in this study: Cohort A will consist of participants with clear cell (cc) RCC and Cohort B will consist of participants with non-clear cell (ncc) RCC.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A (clear cell RCC cohort) participant must have histologically confirmed diagnosis of clear cell RCC or RCC with clear cell component (with or without sarcomatoid features).
* Cohort B (non-clear cell RCC cohort) participant must have histologically confirmed diagnosis of non-clear cell RCC (with or without sarcomatoid features). Participants with tumors that have a component of clear cell histology are not eligible for inclusion in Cohort B.
* Has locally advanced/metastatic disease, i.e., newly diagnosed Stage IV RCC per American Joint Committee on Cancer (AJCC) or have recurrent disease.
* Has measurable disease per RECIST 1.1 as assessed by BICR.
* Has received no prior systemic therapy for advanced RCC. Prior neoadjuvant/adjuvant therapy for RCC is acceptable if completed >12 months prior to allocation.
* Must provide adequate tissue for biomarker analysis for Cohorts A and B from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Participants receiving bone resorptive therapy (including but not limited to bisphosphonate or RANK-L inhibitor) must have therapy initiated at least 2 weeks prior to treatment allocation.
* Has Karnofsky Performance Status (KPS) ≥70%, as assessed within 10 days prior to treatment allocation.
* Demonstrates adequate organ function.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.
* Male participants of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to allocation, has had major surgery within 4 weeks or radiation therapy within 2 weeks prior to allocation, or who has not recovered (i.e., ≤ Grade 1 or to Baseline) from AEs due to prior treatment.
* Had prior treatment with any anti-programmed cell death 1 (anti-PD-1), or anti-programmed cell death ligand 1 (PD-L1), or PD-L2 agent or an antibody targeting any other immune-regulatory receptors or mechanisms. Examples of such antibodies include antibodies against indoleamine-2,3-dioxygenase (IDO), PD-L1, interleukin 2 receptors (IL-2R), glucocorticoid-induced tumor necrosis factor receptor-related protein (GITR).
* Has a diagnosis of immunodeficiency OR is receiving a systemic steroid therapy exceeding 10 mg daily dose of prednisone or equivalent or any other form of immunosuppressive therapy within 7 days prior to allocation, except in the case of central nervous system (CNS) metastases (see below).
* Has an active autoimmune disease requiring systemic treatment within the past 2 years OR a documented history of clinically severe autoimmune disease.
* Has a known additional malignancy that has had progression or has required active treatment in the last 3 years. Note: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, such as breast cancer in situ, that has undergone potentially curative therapy are acceptable.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has known history of Hepatitis B or known active Hepatitis C.
* Has received a live virus vaccine within 30 days of allocation.
* Has had a prior solid organ transplant.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] McDermott DF, Lee JL, Bjarnason GA, Larkin JMG, Gafanov RA, Kochenderfer MD, Jensen NV, Donskov F, Malik J, Poprach A, Tykodi SS, Alonso-Gordoa T, Cho DC, Geertsen PF, Climent Duran MA, DiSimone C, Silverman RK, Perini RF, Schloss C, Atkins MB. Open-Label, Single-Arm Phase II Study of Pembrolizumab Monotherapy as First-Line Therapy in Patients With Advanced Clear Cell Renal Cell Carcinoma. J Clin Oncol. 2021 Mar 20;39(9):1020-1028. doi: 10.1200/JCO.20.02363. Epub 2021 Feb 2. PMID 33529051
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] McDermott DF, Lee JL, Ziobro M, Suarez C, Langiewicz P, Matveev VB, Wiechno P, Gafanov RA, Tomczak P, Pouliot F, Donskov F, Alekseev BY, Shin SJ, Bjarnason GA, Castellano D, Silverman RK, Perini RF, Schloss C, Atkins MB. Open-Label, Single-Arm, Phase II Study of Pembrolizumab Monotherapy as First-Line Therapy in Patients With Advanced Non-Clear Cell Renal Cell Carcinoma. J Clin Oncol. 2021 Mar 20;39(9):1029-1039. doi: 10.1200/JCO.20.02365. Epub 2021 Feb 2. PMID 33529058
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Clear Cell Renal Cell Carcinoma (ccRCC): Participants with ccRCC received pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 doses (approximately 24 months). Eligible participants with ccRCC who experienced disease progression received a second course of up to 17 additional doses of pembrolizumab.
- Cohort B: Non-clear Cell RCC (nccRCC): Participants with nccRCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months). Eligible participants with nccRCC who experienced disease progression received a second course of up to 17 additional doses of pembrolizumab.
Period: Overall Study
Arm/Group | Cohort A: Clear Cell Renal Cell Carcinoma (ccRCC) | Cohort B: Non-clear Cell RCC (nccRCC)
Started | 110 | 165
Received Second Course of Pembrolizumab | 3 | 5
Completed | 0 | 0
Not Completed | 110 | 165
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Participation in Study Terminated by Sponsor | 37 | 48
Not completed — Death | 70 | 112

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: Clear Cell Renal Cell Carcinoma (ccRCC): Participants with ccRCC received pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 doses (approximately 24 months).
- Cohort B: Non-clear Cell RCC (nccRCC): Participants with nccRCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
- Total: Total of all reporting groups
Arm/Group | Cohort A: Clear Cell Renal Cell Carcinoma (ccRCC) | Cohort B: Non-clear Cell RCC (nccRCC) | Total
Number analyzed (Participants) | 110 | 165 | 275
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (11.0) | 60.0 (12.3) | 61.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 56 | 80
  Male | 86 | 109 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 104 | 156 | 260
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 11 | 17 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 98 | 145 | 243
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: Up to approximately 52 months
Population: All allocated participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort A: Clear Cell RCC (ccRCC): Participants with ccRCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell RCC (nccRCC)
Number analyzed (Participants) | 110 | 165
Percentage of Participants | 36.4 [27.4 to 46.1] | 26.7 [20.1 to 34.1]

2. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR with confirmation. The DOR as assessed using RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least one dose of study treatment and had confirmed complete response or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC): Participants with nccRCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 40 | 44
Months | 18.9 [2.3 to NA] — NA=DOR upper limit not reached at time of data cut-off due to insufficient number of responding participants with PD | 29.0 [2.8 to NA] — NA=DOR upper limit not reached at time of data cut-off due to insufficient number of responding participants with PD

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who have achieved CR, PR, or Stable Disease (SD) for at least 6 months based on assessments by the BICR per RECIST 1.1. CR is defined as disappearance of all target lesions, PR is defined as at least a 30% decrease in the sum of diameters of target lesions, SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 110 | 165
Percentage of Participants | 58.2 [48.4 to 67.5] | 43.0 [35.4 to 51.0]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first dose of study treatment to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 110 | 165
Months | 7.1 [5.6 to 11.0] | 4.2 [2.9 to 5.6]

5. Secondary Outcome: Overall Survival
Description: OS was defined as the time from first dose of study treatment to death due to any cause
Time Frame: Up to approximately 66 months
Population: All allocated participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 110 | 165
Months | 40.7 [31.1 to 52.6] | 29.9 [24.3 to 37.4]

6. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure.
Time Frame: Up to approximately 27 months
Population: All allocated participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 110 | 165
Participants | 109 | 155

7. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 6
Time Frame: Up to approximately 24 months
Population: All allocated participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Clear Cell RCC (ccRCC) | Cohort B: Non-clear Cell Renal Cell Carcinoma (nccRCC)
Number analyzed (Participants) | 110 | 165
Participants | 23 | 25

ADVERSE EVENTS:
Time Frame: Up to approximately 66 months
Description: The safety analysis population includes all allocated participants who received at least one dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Therefore, MedDRA preferred terms "Neoplasm Progression", "Malignant Neoplasm Progression" and "Disease Progression" not related to the drug are excluded.
Groups:
- Cohort A: ccRCC First Course: Participants with clear cell RCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
- Cohort B: nccRCC First Course: Participants with non-clear cell RCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months).
- Cohort A: ccRCC Second Course: Participants with clear cell RCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months). Eligible participants with ccRCC who experienced disease progression received up to 17 additional doses of pembrolizumab.
- Cohort B: nccRCC Second Course: Participants with non-clear cell RCC received pembrolizumab 200 mg IV Q3W for up to 35 doses (approximately 24 months). Eligible participants with nccRCC who experienced disease progression received up to 17 additional doses of pembrolizumab.
Arm/Group | Cohort A: ccRCC First Course | Cohort B: nccRCC First Course | Cohort A: ccRCC Second Course | Cohort B: nccRCC Second Course
All-Cause Mortality (participants affected / at risk) | 71/110 | 113/165 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 52/110 | 47/165 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 105/110 | 142/165 | 3/3 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ccRCC First Course (N=110) | Cohort B: nccRCC First Course (N=165) | Cohort A: ccRCC Second Course (N=3) | Cohort B: nccRCC Second Course (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ccRCC First Course (N=110) | Cohort B: nccRCC First Course (N=165) | Cohort A: ccRCC Second Course (N=3) | Cohort B: nccRCC Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 15 (16) | 19 (24) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 11 (11) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 16 (17) | 26 (27) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 22 (28) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (23) | 18 (23) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 35 (58) | 40 (65) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 13 (16) | 15 (18) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 6 (6) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 22 (26) | 28 (38) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 27 (37) | 0 (0) | 0 (0)
Asthenia (General disorders) | 13 (23) | 19 (22) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 7 (7) | 9 (10) | 0 (0) | 0 (0)
Fatigue (General disorders) | 43 (51) | 42 (48) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 10 (24) | 7 (13) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 8 (9) | 14 (16) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 17 (21) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (9) | 11 (16) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (7) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 9 (10) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (15) | 14 (15) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (15) | 15 (17) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 12 (13) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 13 (15) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 19 (23) | 12 (15) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (9) | 5 (11) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (9) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 10 (10) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 22 (24) | 25 (29) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (9) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (9) | 3 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (18) | 7 (10) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (54) | 29 (40) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 22 (28) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 10 (15) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 15 (15) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (13) | 6 (9) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (17) | 18 (24) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 8 (8) | 6 (7) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (13) | 13 (14) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (6) | 6 (9) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 26 (30) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 15 (19) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (11) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (9) | 10 (11) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 41 (54) | 37 (48) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 17 (23) | 19 (24) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (11) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (11) | 11 (12) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT02853344/Prot_SAP_000.pdf